CLINICAL TRIAL: NCT00209833
Title: Protocol for the Treatment of Adults Aged </= 60 Years With De Novo Acute Myeloblastic Leukaemia or Secondary AML or RAEB-T (AML 01/99 Trial)
Brief Title: Treatment of Adults Aged Up to 60 Years With De Novo Acute Myeloblastic Leukaemia,Secondary AML, or RAEB-T
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: University of Ulm (Other); Johann Wolfgang Goethe University Hospital (Other); University Hospital Freiburg (Other); University Hospital Augsburg (Other); Humboldt-Universität zu Berlin (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Ghent (Other); Medizinische Universitätsklinik Tübingen (Unknown); Klinikum Hanover-Siloah Hospital (Other); Ev. Krankenhaus Essen-Werden (Unknown); Klinikum Wuppertal GmbH (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML 01/99 trial
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-11-18 (Estimated); Status verified 2005-09

CONDITIONS: De Novo Akute Myeloid Leukemia (AML); Secondary Acute Myeloid Leukemia (AML); Refractory Anemia With Excess of Blasts in Transformation
MeSH Terms: interventions — Cytarabine; Idarubicin; Etoposide; fludarabine; Granulocyte Colony-Stimulating Factor; Daunorubicin

INTERVENTIONS:
Drug: Cytarabine
Drug: Idarubicin
Drug: Etoposide
Drug: Fludarabine
Drug: G-CSF
Drug: Daunorubicine

SUMMARY:
This randomized phase II/III trial investigates the antileukemic activity and toxicity of the FLAG-Ida regimen as a second induction course in patients with acute myeloid leukaemia and bad response to the first induction cycle and/or with a high risk karyotype and compares the antileukemic activity and toxicity of high dose cytarabine/daunorubicin vs. autologous peripheral blood stem cell transplantation as late consolidation therapy in standard risk patients.

DETAILED DESCRIPTION:
Assessment of the antileukemic activity and toxicity of the FLAG-Ida regimen as a second induction course in patients with bad response to the first induction cycle and/or with a high risk karyotype.

Optimization of the late consolidation therapy in standard risk patients (SR) by a prospective randomized trial comparing a high-dose cytarabine/daunorubicin (HD-Ara-C/DNR) based late consolidation therapy with an autologous peripheral blood stem cell transplantation (PBSCT)

Assessment of the antileukemic activity of the different treatment elements by monitoring residual disease (MRD) after induction, early and late consolidation by Real-time PCR

Assessment of the prognostic relevance of minimal residual disease by quantification of the residual leukemic burden in haematological remission by Real-time PCR during follow-up

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of de-novo AML, FAB M 1, 2, 4 - 7
* diagnosis of secondary AML after chemo-/radiotherapy or MDS
* diagnosis of RAEB-T
* age between 16 and 60 years (including 60 years)
* women after exclusion of pregnancy
* written informed consent

Exclusion Criteria:

* patients with severe disease of the heart (e.g. cardial failure NYHA III/IV; history of myocardial infarction within the last 6 months;severe ventricular arrythmias (Lown III to IV)
* patients with DLCO < 50%
* patients with creatinine clearance < 60 ml/min
* patients with bilirubin > 2mg% (34.2 mmol/L)
* patients with severe complications of the leukaemia such as uncontrolled bleeding, pneumonia with hypoxia or shock
* patients with a psychiatric, addictive, or any disorder which compromises ability to give truly informed consent for participating in this study
* HIV positivity
* patients with a t(15;17) translocation

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 1999-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Efficacy and toxicity of FLAG-Ida as second induction course in high risk patients.
Efficacy and toxicity of high-dose cytarabin/daunorubicin (HD-Ara-C/DNR) based late consolidation therapy vs. autologous peripheral blood stem cell transplantation in standard risk patients.

SECONDARY OUTCOMES:
Monitoring residual disease (MRD) after induction, early and late consolidation by Real-time PCR.
Assessment of the prognostic relevance of minimal residual disease by quantification of minimal residual disease.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Ganser, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Thol F, Bollin R, Gehlhaar M, Walter C, Dugas M, Suchanek KJ, Kirchner A, Huang L, Chaturvedi A, Wichmann M, Wiehlmann L, Shahswar R, Damm F, Gohring G, Schlegelberger B, Schlenk R, Dohner K, Dohner H, Krauter J, Ganser A, Heuser M. Mutations in the cohesin complex in acute myeloid leukemia: clinical and prognostic implications. Blood. 2014 Feb 6;123(6):914-20. doi: 10.1182/blood-2013-07-518746. Epub 2013 Dec 13. PMID 24335498
- [Derived] Buchner T, Schlenk RF, Schaich M, Dohner K, Krahl R, Krauter J, Heil G, Krug U, Sauerland MC, Heinecke A, Spath D, Kramer M, Scholl S, Berdel WE, Hiddemann W, Hoelzer D, Hehlmann R, Hasford J, Hoffmann VS, Dohner H, Ehninger G, Ganser A, Niederwieser DW, Pfirrmann M. Acute Myeloid Leukemia (AML): different treatment strategies versus a common standard arm--combined prospective analysis by the German AML Intergroup. J Clin Oncol. 2012 Oct 10;30(29):3604-10. doi: 10.1200/JCO.2012.42.2907. Epub 2012 Sep 10. PMID 22965967
- [Derived] Thol F, Damm F, Ludeking A, Winschel C, Wagner K, Morgan M, Yun H, Gohring G, Schlegelberger B, Hoelzer D, Lubbert M, Kanz L, Fiedler W, Kirchner H, Heil G, Krauter J, Ganser A, Heuser M. Incidence and prognostic influence of DNMT3A mutations in acute myeloid leukemia. J Clin Oncol. 2011 Jul 20;29(21):2889-96. doi: 10.1200/JCO.2011.35.4894. Epub 2011 Jun 13. PMID 21670448
- [Derived] Damm F, Heuser M, Morgan M, Wagner K, Gorlich K, Grosshennig A, Hamwi I, Thol F, Surdziel E, Fiedler W, Lubbert M, Kanz L, Reuter C, Heil G, Delwel R, Lowenberg B, Valk PJ, Krauter J, Ganser A. Integrative prognostic risk score in acute myeloid leukemia with normal karyotype. Blood. 2011 Apr 28;117(17):4561-8. doi: 10.1182/blood-2010-08-303479. Epub 2011 Mar 3. PMID 21372155
- [Derived] Wagner K, Damm F, Thol F, Gohring G, Gorlich K, Heuser M, Schafer I, Schlegelberger B, Heil G, Ganser A, Krauter J. FLT3-internal tandem duplication and age are the major prognostic factors in patients with relapsed acute myeloid leukemia with normal karyotype. Haematologica. 2011 May;96(5):681-6. doi: 10.3324/haematol.2010.034074. Epub 2011 Jan 17. PMID 21242187
- [Derived] Thol F, Damm F, Wagner K, Gohring G, Schlegelberger B, Hoelzer D, Lubbert M, Heit W, Kanz L, Schlimok G, Raghavachar A, Fiedler W, Kirchner H, Heil G, Heuser M, Krauter J, Ganser A. Prognostic impact of IDH2 mutations in cytogenetically normal acute myeloid leukemia. Blood. 2010 Jul 29;116(4):614-6. doi: 10.1182/blood-2010-03-272146. Epub 2010 Apr 26. PMID 20421455
- See also: Related Info — http://www.kompetenznetz-leukaemie.de/